CLINICAL TRIAL: NCT06004999
Title: Differential Effects of Whole-Body Vibration and Floor Exercises on Muscle Architecture, Functional Performance, and Well-Being in Pre-Frail Seniors: A Randomized Controlled Trial
Brief Title: Effects of Whole Body Vibration in Pre-frail Individuals Over 65 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, FİLİZ TUNA, Assoc. Prof., Trakya University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TÜTF-GOBEAEK 2022/335
Record Dates: First submitted 2023-06-14; First posted 2023-08-22 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pre-frail
Keywords: Whole body vibration; Pre-frail; Anterior thigh muscle thickness; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration group (Experimental): An exercise program organized by the researchers on the vibration platform will be applied to the pre-frail participants in the vibration group. The exercises will be applied 5 days a week for 6 weeks.
  Interventions: Other: Whole body vibration
- Control group (Active Comparator): An exercise program organized by the researchers (same exercise program as the vibration group) will be applied to the pre-frail participants in the control group on a flat surface. The exercises will be applied 5 days a week for 6 weeks.
  Interventions: Other: The exercise program on flat ground without a vibration platform

INTERVENTIONS:
Other: Whole body vibration — All patients will be pedaling for 5 minutes, followed by a warm-up phase with 5 minutes of stretching for the hamstring, gastrocnemius, soleus, and quadriceps muscles.
  Afterward, the following exercise program on the vibration platform will be applied to the 1st group.
  * Lunge,
  * Squat,
  * Deep squat,
  * Wide stance squat,
  * Calves,
  * Deep calves. The exercise time will be 6 minutes in the first week, and the exercise time will be increased in the following weeks, and the total exercise time will continue at 18 minutes in the last week.
  Arms: Vibration group
Other: The exercise program on flat ground without a vibration platform — All patients will be pedaling for 5 minutes, followed by a warm-up phase with 5 minutes of stretching for the hamstring, gastrocnemius, soleus, and quadriceps muscles.
  Afterward, the following exercise program will be applied to the group.
  The exercise program will be applied to the 2nd group (controls) on flat ground without a vibration platform.
  * Lunge,
  * Squat,
  * Deep squat,
  * Wide stance squat,
  * Calves,
  * Deep calves. The exercise time will be 6 minutes in the first week, and the exercise time will be increased in the following weeks, and the total exercise time will continue at 18 minutes in the last week.
  Arms: Control group

SUMMARY:
In this study, individuals aged 65 and over who applied to the physical medicine and rehabilitation outpatient clinic with any complaint will be evaluated in terms of geriatric syndromes. Patients identified as pre-frail will be randomized into the two exercise groups. Exercises of the first group will be performed on the whole body vibration platform and the second will be performed on a flat surface. Before and after the 6-weeks of exercise program; handgrip strength, anterior thigh muscle thickness, body composition, physical performance, mobility, physical activity, balance, kinesiophobia, mood, quality of life, sleep quality, fatigue will be evaluated in both groups. The aim of the study is to show the possible effects of whole body vibration. The results of the study may offer new treatment options that may help prevent the progression of frailty in pre-frail individuals and may guide similar studies.

DETAILED DESCRIPTION:
Frailty is included in geriatric syndromes and is accepted as a precursor of other geriatric syndromes. The elderly who do not meet all the frailty criteria but are at risk are defined as "pre-frail". In many studies %50 of individuals aged 65 and over who appear healthy have been identified at an early stage and their progression to frailty can be reduced or prevented.

Proven treatment approaches for physical frailty include aerobic and resistive exercise. As a result of this study, it is predicted that whole body vibration may be an alternative treatment modality for "pre-frail " individuals who cannot do aerobic and resistive exercises or who are inconvenient to do these exercises.

In the literature, the effect of whole body vibration on muscle strength, balance, physical performance and spasticity in various age groups have been shown. There are no studies showing the effect of whole body vibration in pre-frail individuals and investigating the effect of whole body vibration on anterior thigh muscle thickness. In this study, pre-frail patients will be randomized into exercise groups. 6-week exercise programme is planned to be performed on whole body vibration platform for one group and on flat ground for the other group. The relationship between whole body vibration application and anterior thigh muscle thickness will be examined by measuring the anterior thigh muscle thickness of all participants via ultrasonography (USG). In addition, the relationship between whole body vibration application and body composition, physical performance, balance, kinesiophobia, mood, fatigue, quality of life and sleep will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years and older
2. Those who agreed to participate in the study
3. Groups that have the authority to understand and listen to the questions posed
4. Having no regular exercise habits

Exclusion Criteria:

1. Communication disorder that prevents storytelling and cooperation
2. Serious neurological disease (central nervous system disorders such as paralysis, spinal cord injury, parkinsonism)
3. Advanced cardiovascular disease (decongestive heart failure, recent myocardial infarction)
4. Serious pulmonary disease (COPD exacerbation, acute pulmonary embolism)
5. Physical disability such as lower extremity amputation, surgery
6. Implant (pacemaker, artificial heart valve, stent, hip replacement, knee replacement)
7. Pregnancy
8. Epilepsy
9. Having gallstones, kidney stones, bladder stones
10. Acute inflammation, infection
11. Acute or previous deep vein thrombosis
12. Presence of a history of malignant disease
13. History of fracture in the last 6 months
14. History of lower extremity surgery in the last 12 months
15. Having a regular exercise habit

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Anterior thigh muscle thickness | Change from baseline anterior thigh muscle thickness at second, fourth and sixth weeks of intervention.
  Anterior thigh muscle thickness will be measured in centimeters by ultrasonography.
Lower Extremity Muscle Strength | Change from baseline lower extremity muscle strength at sixth weeks of intervention
  The lower extremities will be evaluated by chair rise test ( also called chair stand test). This test can be used as a proxy for strength of leg muscles (quadriceps muscle group). The chair stand test measures the amount of time needed for a patient to rise five times from a seated position without using his or her arms; the timed chair stand test is a variation that counts how many times a patient can rise and sit in the chair over a 30-second interval.

SECONDARY OUTCOMES:
Hand grip strength | Change from baseline hand grip strength at sixth weeks of intervention
  Hand grip strength is a reliable measurement when standardised methods and calibrated equipment are used, even when there are different assessors or different brands of dynamometers. Hand grip strength will be measured by Jamar Analogue Hand Dynamometer in kilograms.
Skeletal muscle mass index (SMI) | Change from baseline skeletal muscle mass index at sixth weeks of intervention
  Skeletal muscle mass index (SMI) will be measured in kg/m² by dividing the appendicular skeletal muscle mass (kg) by the square of the height (m) using bioelectrical impedance analysis (BIA).
Physical performance | Change from baseline physical performance at sixth weeks of intervention
  The Short Physical Performance Battery (SPPB) is used to determine physical performance. The SPPB is a composite test that includes assessment of walking speed, balance test, and chair rise test.
Mobility | Change from baseline mobility at sixth weeks of intervention
  Mobility will be determined by the timed get-and-go test. The test measures speed during many functional maneuvers such as standing up, walking, turning, and sitting.
Physical activity | Change from baseline physical activity at sixth weeks of intervention
  Physical activity will be assessed using the International Physical Activity Questionnaire - short form (IPAQ). It provides information about time spent walking, moderate- intensity activity, vigorous-intensity activity and sedentary activity.
Balance | Change from baseline balance at sixth weeks of intervention
  Balance will be scored by Berg balance test and Tinetti balance-gait tests. Berg balance test scores balance between 0 to 56 in which higher score means better outcome. Tinetti balance-gait test scores balance between 0 to 9 in which higher score means better outcome.
Kinesiophobia | Change from baseline kinesiophobia at sixth weeks of intervention
  Kinesiophobia will be determined by the Tampa Kinesiophobia Scale. It consists of 17 questions including pain, injury, fear and avoidance parameters related to physical activities.
Mood | Change from baseline mood at sixth weeks of intervention
  Depression will be assessed using Geriatric Depression Scale. This scale consists of 30 questions. A total score of 0-10 means no depression, 11-13 means likely depression, above 14 means definite depression.
Life quality | Change from baseline life quality at sixth weeks of intervention
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, self-reported measure of health. Life quality will be measured by SF-36. In this test every subgroup is scored between 0 to 100 and higher score means better outcome.
Sleep quality | Change from baseline sleep quality at sixth weeks of intervention
  Sleep quality will be determined by The Pittsburgh Sleep Quality Index (PSQI). The scale includes 7 components. Every component is scored between 0 to 3. A total score above 5 is considered poor sleep quality.
Fatigue | Change from baseline fatigue at sixth weeks of intervention
  Fatigue will be evaluated with the fatigue severity scale. The scale includes 9 questions, each of which consists of a score scale of 1-7. The scale determines the fatigue levels of the participants in the last 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Tuna, Principal Investigator — Trakya University
Locations (1):
- Trakya University Medical Faculty, Edirne, Turkey (Türkiye)

REFERENCES:
- [Background] Morley JE, Haren MT, Rolland Y, Kim MJ. Frailty. Med Clin North Am. 2006 Sep;90(5):837-47. doi: 10.1016/j.mcna.2006.05.019. PMID 16962845
- [Background] Dent E, Martin FC, Bergman H, Woo J, Romero-Ortuno R, Walston JD. Management of frailty: opportunities, challenges, and future directions. Lancet. 2019 Oct 12;394(10206):1376-1386. doi: 10.1016/S0140-6736(19)31785-4. PMID 31609229
- [Background] Stania M, Juras G, Slomka K, Chmielewska D, Krol P. The application of whole-body vibration in physiotherapy - A narrative review. Physiol Int. 2016 Jun 1;103(2):133-145. doi: 10.1556/036.103.2016.2.1. PMID 28639859
- [Background] Lam FM, Lau RW, Chung RC, Pang MY. The effect of whole body vibration on balance, mobility and falls in older adults: a systematic review and meta-analysis. Maturitas. 2012 Jul;72(3):206-13. doi: 10.1016/j.maturitas.2012.04.009. Epub 2012 May 18. PMID 22609157
- [Background] Zhang L, Weng C, Liu M, Wang Q, Liu L, He Y. Effect of whole-body vibration exercise on mobility, balance ability and general health status in frail elderly patients: a pilot randomized controlled trial. Clin Rehabil. 2014 Jan;28(1):59-68. doi: 10.1177/0269215513492162. Epub 2013 Jul 17. PMID 23864514
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253